CLINICAL TRIAL: NCT04176419
Title: Investigating the Effect of a Perioperative Analgesia Protocol on Postoperative Opioid Usage and Pain Control in Patients Undergoing Major Head and Neck Cancer Surgery Requiring Microvascular Free Flap Reconstruction
Brief Title: Perioperative Analgesia on Postoperative Opioid Usage and Pain Control in H&N Cancer Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Workforce shortage
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CASE6319
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain Control; Opioid Consumption
Keywords: Head & neck cancer; Microvascular free flap reconstruction
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Ketamine; Lidocaine; Glucose; Acetaminophen; Gabapentin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Perioperative intervention (preoperative acetaminophen, gabapentin, and celecoxib and intraoperative ketamine and lidocaine).
  The Investigational Drug Service will mix and prepare the study medications necessary for each participant. An Investigational Drug Service staff member will deliver the oral medications to the nursing team in the preoperative holding unit and the IV medications to the anesthesia team in the OR unit.
  Interventions: Drug: Ketamine; Drug: Lidocaine; Drug: Acetaminophen; Drug: Gabapentin; Drug: Celecoxib
- Control Group (Placebo Comparator): Perioperative placebo
  Placebo oral drugs will be encapsulated versions provided by the Investigational Drug Service and will appear identical to the interventional oral drugs. Placebo IV infusions will be prepared by Investigational Drug Service as per institutional guidelines and will appear identical to the interventional IV drugs.
  Interventions: Drug: Placebo Ketamine; Drug: Placebo Lidocaine; Drug: Placebo Acetaminophen; Drug: Placebo Gabapentin; Drug: Placebo Celecoxib

INTERVENTIONS:
Drug: Ketamine — 0.25 mg/kg IV bolus before incision, followed by 0.005 mg/kg/minute IV for the remainder of the surgical case excluding the final 30-45 minutes.
  Other Names: Ketamine Hydrochloride; Ketamine Hydrochloride Injection; USP
  Arms: Treatment Group
Drug: Placebo Ketamine — 0.25 mg/kg IV bolus before incision, followed by 0.005 mg/kg/minute IV for the remainder of the surgical case excluding the final 30-45 minutes.
  Arms: Control Group
Drug: Lidocaine — 1.5 mg/kg IV bolus before incision, followed by infusion of 1.5 mg/kg/hour ideal body weight (max 8 hours) during the case
  Other Names: Lidocaine Hydrochloride and 5% dextrose; lidocaine hydrochloride injection
  Arms: Treatment Group
Drug: Placebo Lidocaine — 1.5 mg/kg IV bolus before incision, followed by infusion of 1.5 mg/kg/hour ideal body weight (max 8 hours) during the case
  Arms: Control Group
Drug: Acetaminophen — 1,000 mg orally at time of check-in to the preoperative unit
  Other Names: Paracetamol; Tylenol; N-acetyl-para-aminophenol; APAP
  Arms: Treatment Group
Drug: Placebo Acetaminophen — 1,000 mg orally at time of check-in to the preoperative unit
  Arms: Control Group
Drug: Gabapentin — 600 mg orally at time of check in to the preoperative unit
  Other Names: Neurontin
  Arms: Treatment Group
Drug: Placebo Gabapentin — 600 mg orally at time of check in to the preoperative unit
  Arms: Control Group
Drug: Celecoxib — 200 mg orally at time of check in to the preoperative unit
  Other Names: Celebrex
  Arms: Treatment Group
Drug: Placebo Celecoxib — 200 mg orally at time of check in to the preoperative unit
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine how a non-opioid pain control regimen, administered before and during surgery, will affect postoperative pain control and total opioid consumption in head and neck cancer participants undergoing cancer surgery with free flap reconstruction.

DETAILED DESCRIPTION:
This study will help the study team determine how the experimental, non-opioid pain control regimen affects opioid-related side effects, participant satisfaction with pain management, PACU length of stay, hospital length of stay, chronic pain level, and chronic pain-related disability in participants, and to determine the safety and tolerability of the non-opioid pain control regimen in head and neck cancer patients undergoing cancer surgery with free flap reconstruction. Ketamine, Lidocaine, Acetaminophen, Gabapentin, and Celecoxib are FDA-approved drugs that have been approved for use individually, and have been used in combination for perioperative pain control. However, the use of these five drugs together in head and neck cancer patients undergoing free flap reconstruction has not been studied, which is why this study is experimental.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing head & neck free flap reconstruction at the Cleveland Clinic Main Campus
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergy to lidocaine, ketamine, acetaminophen, gabapentin, and/or celecoxib
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Ketamine, Lidocaine or other agents used in this study
* Subjects receiving any other investigational agents
* Inadequate renal function (serum creatinine ≥ 2 mg/dl) within 30 days
* Inadequate hepatic function (total bilirubin ≥ 2 x the institutional ULN and/or AST or ALT ≥3 x the institutional ULN) within 30 days
* Known or suspected history of illicit drug abuse (including opioids but excluding tobacco and EtOH) within the past 6 months
* Pregnancy
* Contraindication to lidocaine (heart block, heart failure with EF < 30%) as determined by history of Congestive Heart Failure, or as determined by preoperative evaluation for surgical clearance
* In the opinion of the investigator, subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption measured in daily morphine equivalent | at 48 hours postop
  Total opioid consumption measured in daily morphine equivalent
Pain levels on Visual Analog Scale (VAS) | Pre-Op, 24 hours postop, and 48 hours postop
  Change in pain levels on Visual Analog Scale (VAS 0-100mm scale with higher scores corresponding to more pain)

SECONDARY OUTCOMES:
Average Opioid Related Symptom Distress Scale (ORSDS) scores | at 96 hours after surgery, and at discharge (an average of 1 week)
  Average Opioid Related Symptom Distress Scale (ORSDS) scores
  The OR-SDS is used to assess subject-reported levels of severity concerning 12 symptoms known to be associated with opioid medication usage. Symptom frequency, severity, and how bothersome symptom was is rated from 1-4 with higher . The average score for each symptom is calculated by taking the mean of patient-reported score. Total possible severity score: 0 (less severe) to 4 (more severe).
Average Patient satisfaction with pain management scores | at the time of discharge (an average of 1 week)
  Average scores for Internally-developed "patient satisfaction with pain management" questionnaire.
  Domains include pain expected vs experienced, frequency of severe pain, promptness of care team, effectiveness of treatment, and future preferences
  Domain scores range from 1-5 with higher scores mean worse outcomes (more severe pain, poor quality of care)
  Domains are distinct and are not summarized with a "total"score.
Time to first flatulence and defecation | an average of 7 days
  Time to first flatulence and defecation from end of surgical case

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ku, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States